CLINICAL TRIAL: NCT06335459
Title: The Epidemiology and Risk Factors of Hallux Valgus in Upper Egypt
Brief Title: Epidemiology of Bunion and Risk Factors
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hossam Khaled Mohamed Ahmed, The epidemiology and risk factors of Hallux Valgus in upper Egypt, Assiut University
Other Study IDs: Epidemiology of bunion
Record Dates: First submitted 2024-03-15; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Hallux Valgus and Bunion
Keywords: bunion; risk factors; epidemiology; upper egypt
MeSH Terms: conditions — Hallux Valgus; Bunion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: epidemiology — Analysis of 2000 AP WB radiographs of Foot in Upper Egypt For Random People and determind cases of Hallux valgus and calculate the prevalence

SUMMARY:
Analysis of the collected data to determine:

* Prevalence.
* Risk factors. Radiological and clinical patterns and their association with specific risk factors Of Hallux Valgus

DETAILED DESCRIPTION:
Hallux valgus (HV) is a common foot deformity whose multifactorial and complex and associated with other foot deformities. It is a common 1st ray deformity characterized by excessive angulation, rotation, and lateral deviation of the great toe at the first metatarsophalangeal joint . There are many symptoms of HV include poor fitting shoes, plantar foot pain, and pain in the medial first MTP joint .The resultant deformity causes pain and discomfort, which decreases the physical function of the foot and has been identified as a risk factor for falls in older people . Systematic reviews estimated the prevalence of HV to be more frequent with Old age and is more prevalent in women . Several risk factors for HV have been identified HV is associates with wearing high-heeled or narrow shoes . Foot problems are prevalent in old aged and are thought to be associated with high heels and narrow shoes The relationship between HV and obesity is less clear. Some studies have found an association between HV and increasing body mass index whereas others have found no association. Most recently, it has been suggested that the association between HV and BMI differs between the genders, with a lower prevalence with increasing BMI in women but no association in men and in Upper Egypt the principle investigator aim to collect data through a cross sectional study to know the prevalence and calculate the percentage of each certain risk factor through AP Standing Foot and evaluate HV angles and determind who has HV and then calaculate the prevalence and determind associated Risk Factors , while collecting cases the principle investigator focus on Emergency Unit on people without Foot Trauma , no neurological deficit and from outpatient clinic

ELIGIBILITY:
Inclusion Criteria:

* aged (18 - 80) including both sexes Males and Females
* Patients with no Foot trauma or Neurological deficit

Exclusion Criteria:

1. Post traumatic Hallux valgus
2. post infection Hallux valgus
3. Post Surgical Hallux valgus -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: randomly taken people 2000 person taken to do AP - Lateral standing position Foot - sessamoid and full History taken with clinical examination and a Questionnaira about knowledge about bunion and if there is past medical seek for help or not
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-07-24 (Estimated); Primary Completion 2025-04-05 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
History taken and well clinical examination and AP Foot standing position of 2000 randomly case with determination of Hallux Valgus angles knowing if It's Hallux Valgus or not calculating The prevalence | baseline
  Calculate the prevalence of Hallux Valgus by history taken and clinical examination of 2000 cases randomly selected and measuring of Hallux Valgus angles for the participants to know the prevalence

REFERENCES:
- [Background] Hecht PJ, Lin TJ. Hallux valgus. Med Clin North Am. 2014 Mar;98(2):227-32. doi: 10.1016/j.mcna.2013.10.007. Epub 2013 Dec 8. PMID 24559871
- [Background] Steadman J, Barg A, Saltzman CL. First Metatarsal Rotation in Hallux Valgus Deformity. Foot Ankle Int. 2021 Apr;42(4):510-522. doi: 10.1177/1071100721997149. Epub 2021 Mar 25. PMID 33764800
- [Background] Menz HB, Marshall M, Thomas MJ, Rathod-Mistry T, Peat GM, Roddy E. Incidence and Progression of Hallux Valgus: A Prospective Cohort Study. Arthritis Care Res (Hoboken). 2023 Jan;75(1):166-173. doi: 10.1002/acr.24754. Epub 2022 Aug 31. PMID 34268894
- [Background] Menz HB, Roddy E, Marshall M, Thomas MJ, Rathod T, Peat GM, Croft PR. Epidemiology of Shoe Wearing Patterns Over Time in Older Women: Associations With Foot Pain and Hallux Valgus. J Gerontol A Biol Sci Med Sci. 2016 Dec;71(12):1682-1687. doi: 10.1093/gerona/glw004. Epub 2016 Feb 1. PMID 26834078
- [Background] Barnish MS, Barnish J. High-heeled shoes and musculoskeletal injuries: a narrative systematic review. BMJ Open. 2016 Jan 13;6(1):e010053. doi: 10.1136/bmjopen-2015-010053. PMID 26769789